CLINICAL TRIAL: NCT02637141
Title: A Phase 2a, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of AMG 714 in Adult Patients With Celiac Disease
Brief Title: A Study to Evaluate the Efficacy and Safety of AMG 714 in Adult Patients With Celiac Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CELIM-NRCD-001; 2015-003647-19 (EudraCT Number)
Record Dates: First submitted 2015-11-28; First posted 2015-12-22 (Estimated); Results first posted 2019-12-03 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-10

CONDITIONS: Celiac Disease
Keywords: celiac; gluten; Interleukin 15 (IL-15); AMG 714; gluten challenge
MeSH Terms: conditions — Celiac Disease | interventions — AMG-714

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- AMG 714 150 mg (Experimental): Participants received 150 mg AMG 714 via subcutaneous injection once every 2 weeks for a total of 6 doses over 10 weeks from day 0. Participants received gluten-free cookies twice a day for the first 2 weeks and gluten-containing cookies twice a day from weeks 2 to 12 (gluten-challenge).
  Interventions: Biological: AMG 714; Other: Placebo Gluten Challenge; Other: Gluten Challenge
- AMG 714 300 mg (Experimental): Participants received 300 mg AMG 714 via subcutaneous injection once every 2 weeks for a total of 6 doses over 10 weeks from day 0. Participants received gluten-free cookies twice a day for the first 2 weeks and gluten-containing cookies twice a day from weeks 2 to 12 (gluten-challenge).
  Interventions: Biological: AMG 714; Other: Placebo Gluten Challenge; Other: Gluten Challenge
- Placebo (Placebo Comparator): Participants received placebo subcutaneous injection once every 2 weeks for a total of 6 doses over 10 weeks from day 0. Participants received gluten-free cookies twice a day for the first 2 weeks and gluten-containing cookies twice a day from weeks 2 to 12 (gluten-challenge).
  Interventions: Biological: Placebo; Other: Placebo Gluten Challenge; Other: Gluten Challenge

INTERVENTIONS:
Biological: AMG 714 — AMG 714 administered by subcutaneous injection
  Other Names: PRV-015
  Arms: AMG 714 150 mg; AMG 714 300 mg
Biological: Placebo — Matching placebo to AMG 714 administered by subcutaneous injection
  Arms: Placebo
Other: Placebo Gluten Challenge — Gluten-free cookies (Finnish rusks)
Other: Gluten Challenge — Gluten-containing cookies (Finnish rusks), 1-2 g gluten per serving

SUMMARY:
This study is designed to evaluate the efficacy and safety of AMG 714 for the attenuation of the effects of gluten exposure in adult patients with celiac disease during a gluten challenge.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of celiac disease by intestinal biopsy at least 12 months prior to screening
* On a gluten-free diet for at least 12 months
* Negative celiac serology
* Avoidance of pregnancy

Exclusion Criteria:

* Severe complications of celiac disease, such as refractory celiac disease
* Celiac symptoms
* Other concomitant autoimmune disease
* Chronic, active gastrointestinal disease
* Infections, concomitant diseases
* Prohibited medications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-04-13 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2017-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amgen, MD, Study Director — Amgen
Locations (3):
- Finland (3):
  - ODL, Oulu
  - Tampere University Hospital, Tampere
  - CRST, Turku

IPD SHARING:
Plan to Share IPD: Yes
Publication in peer-reviewed journal

REFERENCES:
- [Derived] Lahdeaho ML, Scheinin M, Vuotikka P, Taavela J, Popp A, Laukkarinen J, Koffert J, Koivurova OP, Pesu M, Kivela L, Lovro Z, Keisala J, Isola J, Parnes JR, Leon F, Maki M. Safety and efficacy of AMG 714 in adults with coeliac disease exposed to gluten challenge: a phase 2a, randomised, double-blind, placebo-controlled study. Lancet Gastroenterol Hepatol. 2019 Dec;4(12):948-959. doi: 10.1016/S2468-1253(19)30264-X. Epub 2019 Sep 4. PMID 31494096
- See also: Related Info — http://www.celimmune.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at three sites in Finland.
Pre-assignment Details: Participants who met the study entry criteria were randomized at a 1:1:1 ratio to receive 150 mg or 300 mg AMG 714 or placebo once every 2 weeks for a total of 6 administrations over a period of 10 weeks. Randomization was stratified by study site and sex.
Period: Overall Study
Arm/Group | AMG 714 150 mg | AMG 714 300 mg | Placebo
Started | 22 | 22 | 20
Received Study Drug | 22 | 21 | 19
Completed | 20 | 20 | 19
Not Completed | 2 | 2 | 1
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AMG 714 150 mg | AMG 714 300 mg | Placebo | Total
Number analyzed (Participants) | 22 | 22 | 20 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (15.5) | 47.8 (15.1) | 54.7 (14.9) | 51.0 (15.2)
Age, Customized [Count of Participants; unit: Participants]
  18 - 64 years | 17 | 20 | 12 | 49
  ≥ 65 years | 5 | 2 | 8 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 14 | 47
  Male | 6 | 5 | 6 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 21 | 22 | 20 | 63
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 22 | 22 | 20 | 64
Small Intestinal Villous Height to Crypt Depth Ratio [Mean (Standard Deviation); unit: ratio] — Villi are the small fingerlike projections that line the small intestine and promote nutrient absorption and are often shortened in patients with celiac disease. Crypts are grooves between the villi that are often elongated in patients with celiac disease (crypt hyperplasia). A lower villous height to crypt depth ratio (VH:CD) indicates a flattening of the mucosa and more severe intestinal injury. Population: The per protocol 1 (PP1) population included randomized participants who received at least 1 dose of study drug, were histologically evaluable (provided a post-treatment biopsy samples) and received gluten challenge for at least 1 week.
  ratio
    number analyzed (Participants) | 15 | 19 | 15 | 49
    (all) | 2.12 (0.251) | 2.19 (0.343) | 2.19 (0.426) | 2.17 (0.341)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Villous Height to Crypt Depth Ratio (VH:CD) at Week 12
Description: Attenuation of the effects of gluten exposure was assessed by measuring the percent change from baseline in villous height to crypt depth ratio after 10 weeks of gluten challenge.
  Villi are the small fingerlike projections that line the small intestine and promote nutrient absorption and are often shortened in patients with celiac disease. Crypts are grooves between the villi that are often elongated in patients with celiac disease. A decreased VH:CD ratio indicates worsening disease.
  Small bowel biopsies were performed at baseline and week 12; histological assessments were performed by a blinded central pathologist.
Time Frame: Baseline and week 12
Population: The per protocol 1 (PP1) population included randomized participants who received at least 1 dose of study drug, were histologically evaluable (provided a post-treatment biopsy sample) and received gluten challenge for at least 1 week.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | AMG 714 150 mg | AMG 714 300 mg | Placebo
Number analyzed (Participants) | 15 | 19 | 15
percent change | -62.66 (5.39) | -53.78 (4.83) | -60.17 (5.22)
Statistical Analysis 1: Comparison: AMG 714 150 mg vs Placebo; Test type: Superiority — P-values smaller than 0.05 were considered statistically significant; p = 0.7271, ANCOVA; The model included baseline VH:CD ratio, site, and sex as covariates and treatment group as a fixed effect; LS Mean Difference = -2.49, 95% CI 2-sided [-16.82 to 11.83], Standard Error of Mean 7.10
Statistical Analysis 2: Comparison: AMG 714 300 mg vs Placebo; Test type: Superiority — P-values smaller than 0.05 were considered statistically significant; p = 0.3438, ANCOVA; The model included baseline VH:CD ratio, site, and sex as covariates and treatment group as a fixed effect; LS Mean Difference = 6.39, 95% CI 2-sided [-7.07 to 19.85], Standard Error of Mean 6.67

2. Secondary Outcome: Percent Change From Baseline in Intraepithelial Lymphocyte Density at Week 12
Description: Intraepithelial lymphocytes (IELS) are white blood cells interspersed between epithelial cells of the small and large intestine where they function to preserve the integrity of the mucosal barrier by protecting the epithelium against pathogen or immune-induced pathology. Increased intraepithelial lymphocytes is associated with celiac disease.
  Small bowel biopsies were performed at baseline and week 12; histological assessments were performed by a blinded central pathologist.
Time Frame: Baseline and week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | AMG 714 150 mg | AMG 714 300 mg | Placebo
Number analyzed (Participants) | 15 | 19 | 15
percent change | 95.14 (15.06) | 68.22 (13.64) | 109.46 (14.65)
Statistical Analysis 1: Comparison: AMG 714 150 mg vs Placebo; Test type: Superiority; p = 0.4746, ANCOVA; The model included baseline VH:CD ratio, site, and sex as covariates and treatment group as a fixed effect; LS Mean Difference = -14.32, 95% CI 2-sided [-54.39 to 25.74], Standard Error of Mean 19.85
Statistical Analysis 2: Comparison: AMG 714 300 mg vs Placebo; Test type: Superiority; p = 0.0343, ANCOVA; The model included baseline VH:CD ratio, site, and sex as covariates and treatment group as a fixed effect; LS Mean Difference = -41.24, 95% CI 2-sided [-79.28 to -3.2], Standard Error of Mean 18.85

3. Secondary Outcome: Number of Participants With Improvement in Marsh Score at Week 12
Description: The Marsh classification system describes the stages of damage in the small intestine as seen under a microscope, with possible values of 0, 1, 2, 3a, 3b, or 3c. A score of 0 (best score) indicates that the intestinal lining is normal and celiac disease highly unlikely, a score of 3c (worst score) indicates increased intraepithelial lymphocytes, increased crypt hyperplasia and complete villi atrophy. Improvement is defined as a lower grade on the Marsh score scale compared to baseline.
Time Frame: Baseline and week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AMG 714 150 mg | AMG 714 300 mg | Placebo
Number analyzed (Participants) | 15 | 19 | 15
Participants | 0 | 0 | 0

4. Secondary Outcome: Percent Change From Baseline in Anti-Tissue Transglutaminase (tTG) Immunoglobulin A (IgA) Antibodies at Week 12
Description: Levels of anti-tTG IgA antibodies in serum were determined using an enzyme-linked immunosorbent assay (ELISA) immunoassay.
Time Frame: Baseline and week 12
Population: Per protocol 1 population with available data
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | AMG 714 150 mg | AMG 714 300 mg | Placebo
Number analyzed (Participants) | 15 | 18 | 15
percent change | 5019.77 (1482.59) | 1562.42 (784.83) | 617.53 (866.44)
Statistical Analysis 1: Comparison: AMG 714 150 mg vs AMG 714 300 mg; Test type: Superiority; p = 0.0140, Mixed-effect Model Repeat Measurement; The model included baseline value, treatment group, site, sex, time point, and a time point-by-treatment group interaction term as fixed effects; LS Mean Difference = 4402.25, 95% CI 2-sided [936.39 to 7868.10], Standard Error of Mean 1717.40
Statistical Analysis 2: Comparison: AMG 714 300 mg vs Placebo; Test type: Superiority; p = 0.4228, Mixed-effect Model Repeat Measurement; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = 944.90, 95% CI 2-sided [-1410.65 to 3300.44], Standard Error of Mean 1167.22

5. Secondary Outcome: Change From Baseline in Anti-Deamidated Gliadin Peptide (DGP) Antibodies at Week 12
Description: Levels of serum anti-DGP antibodies (immunoglobulin A [IgA] and immunoglobulin G [IgG]) were determined using ELISA immunoassay.
Time Frame: Baseline and week 12
Population: Per protocol 1 population with available data
Measure: Least Squares Mean (Standard Error); unit: kU/L
Arm/Group | AMG 714 150 mg | AMG 714 300 mg | Placebo
Number analyzed (Participants) | 15 | 18 | 15
kU/L
  Immunoglobulin A | 43.19 (12.85) | 18.47 (10.70) | 25.38 (11.44)
  Immunoglobulin G | 28.29 (21.45) | 17.98 (14.57) | 15.12 (16.02)
Statistical Analysis 1: Comparison: AMG 714 150 mg vs Placebo; Analysis of Change From Baseline in Anti-DGP-IgA; Test type: Superiority; p = 0.3034, Mixed-effect Model Repeat Measurement; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = 17.8, 95% CI 2-sided [-16.68 to 52.29], Standard Error of Mean 17.09
Statistical Analysis 2: Comparison: AMG 714 300 mg vs Placebo; Analysis of Change From Baseline in Anti-DGP-IgA; Test type: Superiority; p = 0.6569, Mixed-effect Model Repeat Measurement; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -6.92, 95% CI 2-sided [-38.11 to 24.28], Standard Error of Mean 15.46
Statistical Analysis 3: Comparison: AMG 714 150 mg vs Placebo; Analysis of Change From Baseline in Anti-DGP-IgG; Test type: Superiority; p = 0.6254, Mixed-effect Model Repeat Measurement; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = 13.17, 95% CI 2-sided [-40.86 to 67.20], Standard Error of Mean 26.77
Statistical Analysis 4: Comparison: AMG 714 300 mg vs Placebo; Analysis of Change From Baseline in Anti-DGP IgG; Test type: Superiority; p = 0.8955, Mixed-effect Model Repeat Measurement; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = 2.86, 95% CI 2-sided [-40.84 to 46.57], Standard Error of Mean 21.66

6. Secondary Outcome: Number of Weekly Bowel Movements at Baseline and Week 12
Description: Participants were asked to record every bowel movement during the study using an electronic diary. If no bowel movements were experienced on any given day, the participant was required to document this using the electronic diary.
Time Frame: Baseline and week 12
Population: Per protocol 1 population with available data
Measure: Mean (Standard Deviation); unit: bowel movements per week
Arm/Group | AMG 714 150 mg | AMG 714 300 mg | Placebo
Number analyzed (Participants) | 15 | 19 | 14
bowel movements per week
  Baseline | 8.9 (3.66) | 10.2 (3.96) | 9.6 (2.92)
  Week 12 | 9.3 (2.58) | 11.5 (5.25) | 11.6 (3.99)
Statistical Analysis 1: Comparison: AMG 714 150 mg vs Placebo; Analysis of Total Weekly Bowel Movements at Week 12; Test type: Superiority; p = 0.1610, Generalized Linear Mixed Model; Generalized linear mixed model with treatment group, site, sex, time (week), and time point-by-treatment group interaction as fixed effects; Ratio of LS Means = 0.83, 95% CI 2-sided [0.63 to 1.08], Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: AMG 714 300 mg vs Placebo; Test type: Superiority; p = 0.7810, Generalized Linear Mixed Model; [statistical method as in outcome 6, analysis 1]; Ratio of LS Means = 1.03, 95% CI 2-sided [0.81 to 1.32], Standard Error of Mean 0.13

7. Secondary Outcome: Number of Participants With Diarrhoea at Baseline and Week 12
Description: The Bristol Stool Form Scale (BSFS) is a pictorial aid to help study participants identify the shape and consistency of their bowel movements. Participants were asked to complete this form daily using an electronic diary at the time of each bowel movement. The BSFS categorizes bowel movements into 7 types, from Type 1 (separate hard lumps, like nuts; hard to pass) to Type 7 (watery, no solid pieces, entirely liquid).
  Diarrhoea was defined as at least one BSFS score >= 6 for the given week.
Time Frame: Baseline and week 12
Population: Per protocol 1 population
Measure: Count of Participants; unit: Participants
Arm/Group | AMG 714 150 mg | AMG 714 300 mg | Placebo
Number analyzed (Participants) | 15 | 19 | 15
Participants
  Baseline | 4 | 9 | 7
  Week 12 | 1 | 5 | 6

8. Secondary Outcome: Percent Change From Baseline in Total Weekly Gastrointestinal Symptom Rating Scale (GSRS) Score at Week 12
Description: The GSRS is a 15-question 7-scale questionnaire used to assess 5 dimensions of gastrointestinal syndromes: diarrhea, indigestion, constipation, abdominal pain, and reflux. Questions are scored between 1 (no discomfort at all) and 7 (very severe discomfort). The total GSRS score is calculated as the sum of the scores of all 15 questions, and ranges from 15 (no discomfort at all) to 105 (very severe discomfort in all 5 dimensions of gastrointestinal syndromes).
Time Frame: Baseline and 12 weeks
Population: Per protocol 1 population with available data
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | AMG 714 150 mg | AMG 714 300 mg | Placebo
Number analyzed (Participants) | 15 | 19 | 14
percent change | 4.14 (9.01) | 14.96 (8.17) | 17.58 (8.93)
Statistical Analysis 1: Comparison: AMG 714 150 mg vs Placebo; Test type: Superiority; p = 0.2761, Mixed-effect Model Repeat Measurement; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -13.44, 95% CI 2-sided [-37.66 to 10.77], Standard Error of Mean 12.33
Statistical Analysis 2: Comparison: AMG 714 300 mg vs Placebo; Test type: Superiority; p = 0.8221, Mixed-effect Model Repeat Measurement; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -2.62, 95% CI 2-sided [-25.51 to 20.27], Standard Error of Mean 11.66

9. Secondary Outcome: Change From Baseline in Total Celiac Disease GSRS (CeD-GSRS) Score at Week 12
Description: The CeD-GSRS score is derived from a subset of questions from the GSRS questionnaire, including the diarrhea, indigestion, and abdominal pain domains (a total of 10 questions), which are each assessed on a scale of 1 (no discomfort at all) to 7 (very severe discomfort).
  The total CeD-GSRS score is calculated as the sum of the scores of all 10 questions, and ranges from 10 (no discomfort at all) to 70 (very severe discomfort in all celiac syndromes).
Time Frame: Baseline and 12 weeks
Population: Per protocol 1 population with available data
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | AMG 714 150 mg | AMG 714 300 mg | Placebo
Number analyzed (Participants) | 15 | 19 | 14
units on a scale | 0.65 (1.52) | 1.77 (1.37) | 3.41 (1.52)
Statistical Analysis 1: Comparison: AMG 714 150 mg vs Placebo; Test type: Superiority; p = 0.1908, Mixed-effect Model Repeat Measurement; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -2.76, 95% CI 2-sided [-6.89 to 1.3], Standard Error of Mean 2.10
Statistical Analysis 2: Comparison: AMG 714 300 mg vs Placebo; Test type: Superiority; p = 0.4088, Mixed-effect Model Repeat Measurement; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -1.64, 95% CI 2-sided [-5.53 to 2.25], Standard Error of Mean 1.98

ADVERSE EVENTS:
Time Frame: From first dose of study drug until week 16
Groups:
- 150 mg AMG 714: Participants received 150 mg AMG 714 via subcutaneous injection once every 2 weeks for a total of 6 doses over 10 weeks from day 0. Participants received gluten-free cookies twice a day for the first 2 weeks and gluten-containing cookies twice a day from weeks 2 to 12 (gluten-challenge).
- 300 mg AMG 714: Participants received 300 mg AMG 714 via subcutaneous injection once every 2 weeks for a total of 6 doses over 10 weeks from day 0. Participants received gluten-free cookies twice a day for the first 2 weeks and gluten-containing cookies twice a day from weeks 2 to 12 (gluten-challenge).
Arm/Group | 150 mg AMG 714 | 300 mg AMG 714 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/21 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21 | 0/19
Other Adverse Events (participants affected / at risk) | 21/22 | 20/21 | 19/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 150 mg AMG 714 (N=22) | 300 mg AMG 714 (N=21) | Placebo (N=19)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 2
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0
Photopsia (Eye disorders) | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 7 | 4 | 6
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 5 | 4
Aphthous ulcer (Gastrointestinal disorders) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 5 | 8 | 6
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 1
Faeces soft (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 3 | 2 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Lip blister (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 7 | 4 | 2
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 1 | 0 | 0
Oral pruritus (Gastrointestinal disorders) | 1 | 0 | 0
Regurgitation (Gastrointestinal disorders) | 0 | 0 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Tongue disorder (Gastrointestinal disorders) | 0 | 1 | 0
Tongue eruption (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 3
Chest pain (General disorders) | 0 | 0 | 2
Chills (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 2 | 5 | 5
Impaired healing (General disorders) | 1 | 0 | 0
Injection site reaction (General disorders) | 8 | 11 | 5
Mucosal dryness (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 2
Conjunctivitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 3 | 2 | 1
Nasopharyngitis (Infections and infestations) | 5 | 7 | 7
Oral herpes (Infections and infestations) | 0 | 2 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 2 | 1
Urinary tract infection (Infections and infestations) | 2 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1 | 0
Procedural headache (Injury, poisoning and procedural complications) | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 1
Blood albumin decreased (Investigations) | 1 | 0 | 0
Blood albumin increased (Investigations) | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1
Blood calcium increased (Investigations) | 0 | 2 | 0
Blood phosphorus increased (Investigations) | 0 | 0 | 1
Blood potassium increased (Investigations) | 0 | 0 | 1
Body temperature decreased (Investigations) | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 1 | 2
Neutrophil count decreased (Investigations) | 0 | 1 | 0
Neutrophil count increased (Investigations) | 1 | 2 | 0
White blood cell count increased (Investigations) | 1 | 3 | 0
White blood cells urine positive (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3 | 3
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 4 | 7 | 8
Migraine (Nervous system disorders) | 1 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Polyneuropathy (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Tonsillolith (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 4 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1 | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Lipoma excision (Surgical and medical procedures) | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 2
Hypertension (Vascular disorders) | 0 | 1 | 0
Temporal arteritis (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2016-08-29): https://cdn.clinicaltrials.gov/large-docs/41/NCT02637141/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-19): https://cdn.clinicaltrials.gov/large-docs/41/NCT02637141/SAP_001.pdf